CLINICAL TRIAL: NCT01391806
Title: The Impact of Preoperative Breast MRI in Newly Diagnosed Breast Cancer. A Prospective Study of Treatment Outcome in Patients Selected for Breast Conserving Surgery in a Norwegian Multidisciplinary Breast Cancer Clinic.
Brief Title: The Impact of Preoperative Breast MRI in Patients With Breast Cancer Selected for Breast Conserving Surgery
Status: Completed | Type: Observational
Sponsor: Nordlandssykehuset HF (Other)
Responsible Party: Toril Rabben/MD DDS PhD Associate professor, Dep. of Surgery, Nordlandssykehuset Bodø, 8092 Bodø and Faculty of Health Sciences, University of Tromsø, 9037 Tromsø, Norway
Other Study IDs: PreopMR 2011
Record Dates: First submitted 2011-07-11; First posted 2011-07-12 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2009-01

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Preoperative breast MRI; Breast-conserving surgery; Mastectomy; Prospective study
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast cancer: Patients selected for breast-conserving surgery based on conventional radiological methods, following the criteria recommended by the Norwegian Breast Cancer Group

SUMMARY:
The purpose of this prospective observational study is to evaluate the impact of preoperative breast MRI in patients with breast cancer selected for breast- conserving surgery. MRI is a more sensitive radiological modality than mammography and ultrasonography. Patients with small breast cancers are, based on conventional modalities, selected for breast-conserving surgery. If preoperative breast MRI reveal additional lesions in the breasts, and malignancy is confirmed histopathologically, this finding leads to a change of surgical method to mastectomy.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the impact of preoperative breast MRI on primary surgical treatment in a highly specialized multidisciplinary breast cancer clinic. The clinic serves a population of 237.000. The diagnostic tools routinely used are conventional mammography, ultrasound with core needle biopsy, and clinical examination including palpation of breast and axillary nodes. If indicated, the examination includes ultrasound examination and fine needle biopsy of axillary glands. We offer all patients selected for breast-conserving surgery preoperative breast MRI.

We include consecutively breast cancer lesions in women aged 35-75 in a prospective study, collecting data from January 2009 to December 2010. The patients are all selected for breast-conserving surgery based on the criteria recommended by the Norwegian Breast Cancer Group. That is, tumor ≤ 4 cm, or acceptable tumor:breast ratio, and age > 35. Multifocal lesions, defined as more than one tumor > 1 cm apart, size of tumor > 4 cm, or a large tumor:breast ratio, extensive ductal carcinoma in situ (DCIS), or known genetic disposition for breast cancer, indicates mastectomy according to these criterias. In addition, when postoperative radiation therapy is contraindicated, mastectomy is indicated. If the patients fill the criteria for breast-conserving surgery, they are offered preoperative breast MRI and included in the study. Patients who either choose mastectomy, or does not get a breast MRI for technical reasons, are excluded from the study. Two experienced breast radiologists evaluate the breast MRIs, and three experienced breast radiologists study the mammographies and perform the ultrasound examinations and biopsies. All additional MRI findings are examined by ultrasound-guided biopsy and given a histological diagnose before it influence the surgical method.

A formal application has been presented to the regional ethical commitee. Since this is an observational study of established practice, the commitee replied that approval was not required.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 35 years and ≤ 75 years
* Indication for breast-conserving surgery according to criteria recommended by the Norwegian Breast Cancer Group:
* Tumor < 4 cm and acceptable tumor:breast ratio
* Tumor not infiltrating skin or pectoral fascia
* No multifocality (that is 2 foci or more, > 1 cm apart)

Exclusion Criteria:

* Patient choose mastectomy
* Technical problems with the MR machine
* Pacemaker
* Anxiety/claustrophobia

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are selected from screening or they are referred to the Breast Diagnostic Clinic for clinical symptoms. The clinic serves a population of 237.000 in Nordland county, Norway. Patients selected for breast-conserving surgery based on conventional radiological examination, that is bilateral mammography and ultrasonography with biopsy, are consecutively included in the study and offered preoperative breast MRI.
Sampling Method: Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Change of surgical method after preoperative breast MRI in breast cancer | Two years of data collection

CONTACTS AND LOCATIONS:
Overall Officials: Toril Rabben, MD DDS PhD, Principal Investigator — Dep. of Surgery, Nordlandssykehuset Bodø, 8092 Bodø, Norway
Locations (1):
- Breast Diagnostic Centre, Dep. of Surgery, Nordlandssykehuset Bodø, Bodø, Norway

REFERENCES:
- See also: Sponsor´s web-site — http://nordlandssykehuset.no